CLINICAL TRIAL: NCT04868682
Title: Addressing Insufficient Positive Airway Pressure Use Among Older Veterans With Obstructive Sleep Apnea
Brief Title: Addressing Insufficient PAP Use in Older Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 20-046
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; positive airway pressure
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the participant or staff who conduct the follow-up assessments will be aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAP Adherence Program (Experimental): Manual-based behavioral treatment to improve PAP adherence and sleep.
  Interventions: Behavioral: PAP Adherence Program
- Active Control (Active Comparator): Manual-based general sleep education program.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: PAP Adherence Program — Manual-based treatment focused on PAP adherence with behavioral strategies to improve PAP adherence and sleep. The intervention involves five individual virtual sessions provided by allied health personnel, with brief monthly telephone contact for up to 6 months. Allied health personnel have regular supervision with a behavioral sleep medicine psychologist.
  Arms: PAP Adherence Program
Behavioral: Active Control — Manual-based general sleep education program. The active control involves five individual virtual sessions provided by allied health personnel, with brief monthly telephone contact for up to 6 months. Allied health personnel have regular supervision with a study clinician.
  Arms: Active Control

SUMMARY:
Obstructive sleep apnea (OSA) is a common problem among middle-aged and older Veterans that is associated with poor nighttime sleep, more daytime sleepiness, poor functioning and worse quality of life. The recommended therapy for most patients with OSA is positive airway pressure (PAP) therapy; however, over time many patients prescribed PAP therapy no longer use it regularly. This study will test the effects of an behavioral treatment specifically designed for middle-aged and older Veterans who have stopped using their PAP device, or are not using it regularly.

Eligible Veterans who are enrolled into the study will receive a baseline assessment that includes questionnaires about sleep, health, and quality of life. After completing the baseline assessment, participants will be randomly assigned to one of two groups. Both groups will meet individually with a "sleep coach" for 5 session over 8 weeks, then they will be contacted by the sleep coach monthly by telephone for up to 6 months. Participants will complete follow-up assessments immediately after the fifth education session and again at 6-months and 12-months.

If successful, this approach has the potential to improve sleep, function and quality of life in middle-aged and older Veterans with OSA.

DETAILED DESCRIPTION:
Background: The most frequently diagnosed sleep disorder among middle-aged and older Veterans is obstructive sleep apnea (OSA), which is associated with serious adverse effects on health, quality of life and survival. Positive airway pressure (PAP) is recommended as first-line treatment (particularly for moderate to severe OSA), but sustained use is difficult to achieve, including among middle-aged and older Veterans, and nearly half of patients with OSA who begin PAP therapy discontinue use within a year.

Significance/Impact: Although OSA is a chronic condition, research to date has primarily focused on increasing initial PAP use in patients with newly diagnosed OSA. In addition, most research has not addressed PAP use in older adults, which is unfortunate given the high prevalence and important adverse effects of OSA on their health and well-being. Prior work suggests that behavioral interventions are effective in improving initial PAP use, but little is known of how to address insufficient PAP use over time.

Innovation: To address this problem, the investigators developed and pilot-tested a structured, manual-based behavioral treatment to address insufficient PAP use among middle-aged and older adults with previously diagnosed OSA. The intervention (5 individual virtual sessions over 8 weeks, then monthly brief telephone contact for up to 6 months) is designed so it can be provided by individuals ("sleep coaches") from various disciplines (supervised remotely by a psychologist) in a variety of settings for maximal implementation.

Specific Aims: Primary Aim 1 will test the efficacy of this intervention for improving PAP usage among middle-aged and older Veterans with previously diagnosed moderate or severe OSA who have insufficient PAP use. The hypotheses are that the intervention will increase objectively measured PAP use over 6-months follow-up, with effects sustained over 12 months. Secondary Aim 2 will test for effects on sleep quality, daytime sleepiness and sleep-related function; and Exploratory Aim 3 will test for effects on health-related quality of life. The hypotheses are that these outcomes will also improve at 6 months, and effects will be sustained at 12 months.

Methodology: The investigators are conducting a randomized, controlled trial to test this new intervention in middle-aged and older Veterans (N=106) with previously diagnosed OSA (moderate or severe) who were prescribed PAP, but have insufficient PAP use (defined as no PAP use over the prior 30 days). Participants will be randomized to one of two groups. Structured assessments at baseline, post-treatment (after session 5) and 6- and 12-months follow-up include objectively measured PAP use (via remote telemonitoring), sleep quality, daytime sleepiness, sleep-related function and health-related quality of life. The investigators will also collect participant experiences and attitudes related to the intervention, and implementation outcome measures (e.g., acceptability, appropriateness, fidelity and staff time as an estimate of cost) to inform future implementation.

Implementation/Next Steps: The long-term goal of this work is to effectively address insufficient PAP use among middle-aged and older Veterans with OSA to improve their sleep and quality of life. If successful, the investigators will develop an implementation package to promote wider implementation of this model of care into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe obstructive sleep apnea (apnea hypopnea index [AHI] > or = 15)
* Previously prescribed positive airway pressure (PAP) therapy
* Insufficient PAP use (defined as no PAP use over the past 30 days)

Exclusion Criteria:

* Severe psychopathology (e.g., active psychosis) that precludes participation in the study
* Severe unstable medical illness that precludes participation in the study
* Significant cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy A. Alessi, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PAP Adherence Program: Manual-based program provided by supervised allied health personnel focused on PAP adherence with behavioral strategies to improve PAP adherence and sleep.
- Active Control: Manual-based general sleep education program provided by supervised allied health personnel.
Period: Post-treatment
Arm/Group | PAP Adherence Program | Active Control
Started | 53 | 53
Completed | 51 | 50
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — 1 refused assessment; 1 in residing in a nursing home; 1 assessment was missed by staff | 1 | 2
Period: Six-month Assessment
Arm/Group | PAP Adherence Program | Active Control
Started | 53 (We attempted to collect 6-month data from all 53 participants in this group. Some participants who did not complete the post-treatment were able to complete the 6-month follow-up.) | 53 (We attempted to collect 6-month data from all 53 participants in this group. Some participants who did not complete the post-treatment were able to complete the 6-month follow-up.)
Completed | 51 | 52
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — Refused | 0 | 1
Period: 12-month Assessment
Arm/Group | PAP Adherence Program | Active Control
Started | 52 (We attempted to collect 12-month data from all 52 surviving participants in this group. Some participants who did not complete the 6-month follow-up were able to complete the 12-month follow-up.) | 53 (We attempted to collect 12-month data from all 53 participants in this group. Some participants who did not complete the 6-month follow-up were able to complete the 12-month follow-up.)
Completed | 50 | 51
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PAP Adherence Program | Active Control | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.7) | 65.5 (9.1) | 66.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 46 | 48 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 16 | 25
  Not Hispanic or Latino | 44 | 37 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 21 | 17 | 38
  White | 22 | 25 | 47
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 3 | 4 | 7
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 21. Higher scores indicate worse outcome.
  units on a scale | 10.4 (4.5) | 9.9 (4.1) | 10.2 (4.3)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — Score range from 0-24. Higher scores indicate worse outcome.
  units on a scale | 9.5 (5.4) | 8.3 (4.9) | 8.9 (5.2)
Functional Outcomes of Sleep Questionnaire-10 items [Mean (Standard Deviation); unit: units on a scale] — Scores range from 5-20. Lower scores indicate worse outcome.
  units on a scale | 14.0 (3.5) | 14.9 (3.7) | 14.4 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: PAP Adherence
Description: Mean hours of PAP use per night calculated for nights 1 to 180 (night 1 is the first night after randomization). Higher numbers indicate a better outcome.
Time Frame: Nights 1 to 180 following randomization
Measure: Mean (Standard Error); unit: hours per night
Arm/Group | PAP Adherence Program | Active Control
Number analyzed (Participants) | 53 | 53
hours per night | 2.16 (0.26) | 0.87 (0.19)
Statistical Analysis 1: Comparison: PAP Adherence Program vs Active Control; Test type: Superiority; p = .0001, t-test, 2 sided; Mean Difference (Final Values) = 1.28, 95% CI 2-sided [0.65 to 1.91], Standard Error of Mean 0.32 — The parameter estimate is the difference in means (treatment vs. control) during the first 180 nights following randomization

2. Secondary Outcome: Sleep Quality
Description: Total score on the Pittsburgh Sleep Quality Index will be used as a measure of sleep quality. Scores range from 0 to 21. Higher scores indicate worse outcome.
Time Frame: 6 months following randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PAP Adherence Program | Active Control
Number analyzed (Participants) | 53 | 53
score on a scale | 7.72 (0.60) | 8.01 (0.59)
Statistical Analysis 1: Comparison: PAP Adherence Program vs Active Control; Test type: Superiority; p = 0.378, Mixed Models Analysis; Mean Difference (Net) = -0.71, 95% CI 2-sided [-2.29 to 0.87], Standard Error of Mean 0.81 — The parameter estimate is the improvement in the outcome from baseline to 6-months for the treatment group versus the same improvement in respect to the control group

3. Secondary Outcome: Daytime Sleepiness
Description: Total score on the Epworth Sleepiness Scale will be used as a measure of daytime sleepiness. Score range from 0-24. Higher scores indicate worse outcome.
Time Frame: 6 months following randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PAP Adherence Program | Active Control
Number analyzed (Participants) | 53 | 53
score on a scale | 6.11 (0.67) | 7.59 (0.67)
Statistical Analysis 1: Comparison: PAP Adherence Program vs Active Control; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -2.78, 95% CI 2-sided [-4.09 to -1.27], Standard Error of Mean 0.72 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Sleep-related Function
Description: Total score on the Functional Outcomes of Sleep Questionnaire (FOSQ-10) will be used as a measure of sleep-related function. Scores range from 5-20. Lower scores indicate worse outcome.
Time Frame: 6 months following randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PAP Adherence Program | Active Control
Number analyzed (Participants) | 53 | 53
score on a scale | 14.65 (0.50) | 15.67 (0.50)
Statistical Analysis 1: Comparison: PAP Adherence Program vs Active Control; Test type: Superiority; p = 0.865, Mixed Models Analysis; Median Difference (Net) = -0.11, 95% CI 2-sided [-1.40 to 1.18], Standard Error of Mean 0.66 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: One year following randomization.
Arm/Group | PAP Adherence Program | Active Control
All-Cause Mortality (participants affected / at risk) | 1/53 | 1/53
Serious Adverse Events (participants affected / at risk) | 6/53 | 1/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP Adherence Program (N=53) | Active Control (N=53)
Mental health distress (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization (Infections and infestations) | 3 (6) | 0 (0)
Hospitalization (Cardiac disorders) | 2 (2) | 1 (1)
Hospitalization (General disorders) | 1 (1) | 0 (0)
Hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT04868682/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT04868682/ICF_000.pdf